CLINICAL TRIAL: NCT05202327
Title: A Phase II Tolerability and Efficacy Study of PDC-1421 Treatment in Adult Patients With Attention-Deficit Hyperactivity Disorder (ADHD), Part II
Brief Title: PDC-1421 Treatment in Adult Patients With ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioLite, Inc. (Industry)
Collaborators: ABVC BioPharma, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLI-1008-002
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Attention-Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Starch

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of three groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Two placebo capsules thrice daily for 56 days (8 weeks).
  Interventions: Drug: Placebo
- Low-dose (Experimental): One placebo capsule and 1 PDC-1421 Capsule, thrice daily for 56 days (8 weeks).
  Interventions: Drug: PDC-1421 Capsule; Drug: Placebo
- High-dose (Experimental): Two PDC-1421 Capsules thrice daily for 56 days (8 weeks).
  Interventions: Drug: PDC-1421 Capsule

INTERVENTIONS:
Drug: PDC-1421 Capsule — PDC-1421 Capsule is a botanical investigational new drug containing the extract of Radix Polygalae (Polygala tenuifolia Willd.) as the active ingredient.
  Other Names: Extract of Radix Polygalae
  Arms: High-dose; Low-dose
Drug: Placebo — The placebo contained corn starch.
  Other Names: Corn Starch
  Arms: Low-dose; Placebo

SUMMARY:
Part II is a double-blind, randomized, parallel-group, placebo-controlled study. The primary objective of this trial is to determine the effective doses and treatment period of PDC-1421 Capsule in subjects with ADHD. The secondary objective is to evaluate the safety of PDC-1421 Capsule in subjects receiving PDC-1421 at various dose levels.

DETAILED DESCRIPTION:
The screening phase is intended for diagnosing and assessing the patient for possible inclusion in the study and for providing an adequate washout period.

At the first stage, a number of 69 subjects will be randomly assigned on a 1:1:1 basis to one of the three arms (1 PDC-1421 Capsule plus 1 placebo TID, 2 PDC-1421 Capsules TID, 2 placebo TID) for 8 weeks and evaluated the safety and efficacy every two weeks during the treatment period. An interim analysis will be conducted to evaluate the efficacy of PDC-1421 and to decide whether it is necessary to enter the second stage of the Part II study in which 30 subjects will be randomly assigned on a 1:1:1 basis to one of the three treatment arms and receive the same treatment.

Simple descriptive statistics with a 95% confidence interval will be performed with data collected in this study wherever applicable. The safety and efficacy data will be analyzed using the non-parametric method wherever appropriate.

The primary endpoint will be analyzed by chi-square test, while the secondary endpoints will be analyzed using the ANOVA or Kruskal-Wallis non-parametric ANOVA test for continuous endpoints and chi-square test for binary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years
2. Female subjects of child-bearing potential must test negative to pregnancy and use appropriate birth control method from the beginning of study to the 15 days later after ending of study
3. Subjects must be able to understand and willing to sign informed consent
4. Able to discontinue the use of any psychotropic medications for the treatment of ADHD symptoms at screening
5. Meet strict operational criteria for adult ADHD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5)
6. A total score of 28 or higher of ADHD Rating Scale-Investigator Rated (ADHD-RS-IV) at screening
7. Have a moderate or severe symptom of ADHD with score of 4 or higher in Clinical Global Impression- Severity (CGI-S) at screening

Exclusion Criteria:

1. Have any clinically significant concurrent medical condition (endocrine, renal, respiratory, cardiovascular, hematological, immunological, cerebrovascular, neurological, anorexia, obesity or malignancy) that has become unstable and may interfere with the interpretation of safety and efficacy evaluations
2. Have any clinically significant abnormal laboratory, vital sign, physical examination, or electrocardiogram (ECG) findings at screening that, in the opinion of the investigator, may interfere with the interpretation of safety or efficacy evaluations
3. Have known serological evidence of human immunodeficiency virus (HIV) antibody
4. Are pregnant as confirmed by a positive pregnancy test at screening
5. Have QTc values >450 msec at screening using Fridericia's QTc formula
6. Have current of bipolar and psychotic disorders
7. Have a current major depression disorder, obsessive-compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder, panic disorder and eating disorder (also if treated but not currently symptomatic) NOTE: Comorbid diagnoses identified during screening and baseline are acceptable provided that ADHD is the primary diagnosis and the comorbid diagnoses will not confound study data or impair subject's ability to participate (per the Investigator's judgement and documented in source note).
8. Have any history of a significant suicide attempt, or possess a current risk of attempting suicide, in the investigator's opinion, based on clinical interview and responses provided on the Columbia-Suicide Severity Rating Scale (C-SSRS).
9. Have a history of jailing or imprisonment in the past 6 months due to worsening of symptoms of ADHD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Improvement ≥ 40% in ADHD-RS-IV From Baseline up to 8 Weeks Treatment | 8 weeks
  The ADHD-RS-IV with Adult Prompts is an 18-item scale based on the DSM-IV-TR criteria for ADHD that provides a rating of the severity of symptoms. The adult prompts serve as a guide to explore more fully the extent and severity of ADHD symptoms and create a framework to ascertain impairment. The odd-numbered 9 items assess inattentive symptoms and the even-numbered 9 items assess hyperactive-impulsive symptoms. Scoring is based on a 4-point, yielding a possible total score of 0-54. Likert-type severity scale: 0 = Never or Rarely, 1 = Sometimes, 2 = Often, 3 = Very Often. Clinicians should score the highest score that is generated for the prompts for each item. The ADHD-RS-IV was assessed from Visit 1 to Visit 7 by the investigator.

SECONDARY OUTCOMES:
Change From Baseline up to 8 Weeks Treatment in the Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version (CAARS-S:S) 5 Subscales T-score. | 8 weeks
  Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version (CAARS-S:S) consists of 26 items rated from 0=not at all, never to 3=very much, very frequently. Four subscales each composed of 5 items (A: inattention/memory problems; B: hyperactivity/restlessness; C: impulsivity/emotional lability; and D: problems with self-concept) as well as a 12-item ADHD index can be computed. The raw scores were converted into standard T-scores by the SAS program which was designed according to the Profile form of CAARS Quik Score forms. The higher T-scores represent a better or worse outcome. A T-score is a standard score with a mean of 50 and a standard deviation of 10 in all samples and across all scales
Change From Baseline up to 8 Weeks in the Sluggish Cognitive Tempo (K-SCT) Score. | 8 weeks
  The K-SCT rating scale queries 15 Sluggish Cognitive Tempo symptoms rated from 0 = Never or Rarely, 1 = Sometimes, 2 = Often, 3 = Very Often, grouped into latent factors of daydreaming, working memory problems, and subjective sleepiness/tiredness. The range for the Total Score is 0-45. The higher values represent a worse outcome for the total score and subscore.
Change From Baseline up to 8 Weeks in the ADHD-RS-IV Inattention Subscale, Hyperactivity-impulsivity Subscale, and Total Scale Raw Score. | 8 weeks
  The ADHD-RS-IV with Adult Prompts is an 18-item scale base on the DSM-IV-TR criteria for ADHD that provides a rating of the severity of symptoms. The adult prompts serve as a guide to explore more fully the extent and severity of ADHD symptoms and create a framework to ascertain impairment. The odd-numbered 9 items assess inattentive symptoms and the even-numbered 9 items assess hyperactive-impulsive symptoms. Scoring is based on a 4-point, yielding a possible summed "total score" of 0-54, "inattentive subscore" of 0-27, and "hyperactive-impulsive subscore" of 0-27. The higher values represent a worse outcome for the total score and subscore. Likert-type severity scale: 0 = Never or Rarely, 1 = Sometimes, 2 = Often, 3 = Very Often.
Number of Participants With Symptom Remission in ADHD-RS-IV From Baseline up to 8 Weeks Treatment | 8 weeks
  The ADHD-RS-IV with Adult Prompts is an 18-item scale base on the DSM-IV-TR criteria for ADHD that provides a rating of the severity of symptoms. The adult prompts serve as a guide to explore more fully the extent and severity of ADHD symptoms and create a framework to ascertain impairment. The odd-numbered 9 items assess inattentive symptoms and the even-numbered 9 items assess hyperactive-impulsive symptoms. Scoring is based on a 4-point, yielding a possible summed "total score" of 0-54, "inattentive subscore" of 0-27, and "hyperactive-impulsive subscore" of 0-27. The higher values represent a worse outcome for the total score and subscore. Likert-type severity scale: 0 = Never or Rarely, 1 = Sometimes, 2 = Often, 3 = Very Often.
Number of Participants With a CGI Score of 2 or Lower From Baseline up to 8 Weeks Treatment | 8 weeks
  Clinical Global Impression-Severity (CGI-S) and Clinical Global Impression-Improvement (CGI-I) score of 2 or lower. The CGI-S is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). CGI-I scores range from 1 (very much improved) through to 7 (very much worse).

CONTACTS AND LOCATIONS:
Locations (6):
- University of California, San Francisco, San Francisco, California, United States
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - Taipei veterans General Hospital, Taipei
  - Linkou chang Gung Memorial Hospital, Taoyuan District